CLINICAL TRIAL: NCT00902486
Title: A Randomized, Double-blind, Placebo Controlled, Dose Ranging, Parallel Group, Phase 2 Study of INCB028050 Compared to Background Therapy in Patients With Active RA With Inadequate Response to Any Disease Modifying Anti-Rheumatic Drugs (DMARD) Therapy Including Biologics
Brief Title: INCB028050 Compared to Background Therapy in Patients With Active Rheumatoid Arthritis (RA) With Inadequate Response to Disease Modifying Anti-Rheumatic Drugs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCB 28050-201
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Results first posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- INCB028050 4 mg QD (Experimental): INCB028050 4mg Once daily (QD)
  Interventions: Drug: INCB028050
- INCB028050 7 mg QD (Experimental): INCB028050 7mg QD
  Interventions: Drug: INCB028050
- INCB028050 10 mg QD (Experimental): INCB028050 10mg QD
  Interventions: Drug: INCB028050
- Placebo (Placebo Comparator): Placebo group may 'cross-over' following 3 months of treatment to receive either active arm #2 (7mg QD) or active arm #3 (10mg QD) of INCB028050 capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INCB028050 — 4 mg capsules QD
  Other Names: Baricitinib
  Arms: INCB028050 4 mg QD
Drug: INCB028050 — 7 mg capsules QD
  Other Names: Baricitinib
  Arms: INCB028050 7 mg QD
Drug: INCB028050 — 10 mg capsule QD
  Other Names: Baricitinib
  Arms: INCB028050 10 mg QD
Drug: Placebo — Placebo matching INCB028050 QD
  Arms: Placebo

SUMMARY:
This was a randomized, double blind, placebo controlled, dose ranging, parallel group study. Participants who had active rheumatoid arthritis (RA) who had inadequate response to any disease modifying anti-rheumatic drug (DMARD) therapy including biologics were enrolled. Screening evaluations were performed within approximately 28 days of randomization. The duration of the study was 6 months with the primary endpoint assessed at 3 months. Eligible participants were randomly assigned to one of three doses (4, 7 or 10 mg QD) of INCB028050 (Baricitinib) or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Must have rheumatoid arthritis which has been inadequately controlled with at least one DMARD
* For subjects receiving antimalarials, they must be treated with antimalarials for at least 6 months and receiving a stable daily dose
* For subjects receiving sulfasalazine, they must be treated with Sulfasalazine (SSZ) for at least 6 months and receiving a stable daily dose of no more than 3 grams per day
* For subjects on methotrexate, they must be treated with methotrexate for at least 6 months, and receiving a stable weekly dose of methotrexate between 7.5 and 25 mg
* For subjects on leflunomide, they must be treated with leflunomide for at least 6 months, and receiving a stable dose of leflunomide between 10 to 20 mg
* For subjects receiving corticosteroids, they must be on a dose not to exceed 10 mg of prednisone daily
* Active rheumatoid arthritis at the time of screening defined by the following: 6 or more joints tender or painful on motion and 4 or more swollen joints and at least one of the following two: Erythrocyte sedimentation rate (ESR) greater than or equal to 28 mm/hr or C-reactive protein (CRP) greater than or equal to 7 mg/liter
* Have evidence of lack of risk for tuberculosis

Exclusion Criteria:

* Current or recent viral, bacterial, fungal, parasitic or mycobacterial infection requiring systemic therapy
* History of infected joint prosthesis
* Subjects who have a current or recent history of severe, progressive, uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary, cardiac, neurological or cerebral disease
* Subjects who have received treatment with the following drugs or drug classes within the specified timeframe: prior treatment with rituximab within 12 months, prior treatment with an oral Janus kinase (JAK) inhibitor, DMARDs or other anti-rheumatic therapies not specified and allowed according to protocol, treatment with any investigational medication within 12 weeks or 5 half-lives (whichever is longer), and treatment with a biologic agent within 12 weeks prior to the first dose of study medication
* Subjects with a past history of neutropenia, thrombocytopenia or anemia requiring transfusion other than at the time of trauma or surgery, and subjects that meet protocol specified laboratory measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2009-05; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (49):
- United States (41):
  - Birmingham, Alabama
  - Paradise Valley, Arizona
  - Peoria, Arizona
  - Phoenix, Arizona
  - Palm Desert, California
  - Santa Maria, California
  - Santa Monica, California
  - Westlake Village, California
  - Whittier, California
  - Denver, Colorado
  - Aventura, Florida
  - Daytona Beach, Florida
  - Gainesville, Florida
  - Lake Mary, Florida
  - Naples, Florida
  - Palm Harbor, Florida
  - Sarasota, Florida
  - Springfield, Illinois
  - South Bend, Indiana
  - Wichita, Kansas
  - Lexington, Kentucky
  - Frederick, Maryland
  - Wheaton, Maryland
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Reno, Nevada
  - Freehold, New Jersey
  - Lake Success, New York
  - Syracuse, New York
  - Charlotte, North Carolina
  - Hickory, North Carolina
  - Middleburg Heights, Ohio
  - Toledo, Ohio
  - Tulsa, Oklahoma
  - Duncansville, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Sellersville, Pennsylvania
  - Houston, Texas
  - San Antonio, Texas
  - Arlington, Virginia
  - Spokane, Washington
- Czechia (8):
  - Brno
  - Chomutov
  - Česká Lípa
  - Hlučín
  - Hustopeče
  - Kroměříž
  - Prague
  - Zlín

REFERENCES:
- [Derived] Taylor PC, Takeuchi T, Burmester GR, Durez P, Smolen JS, Deberdt W, Issa M, Terres JR, Bello N, Winthrop KL. Safety of baricitinib for the treatment of rheumatoid arthritis over a median of 4.6 and up to 9.3 years of treatment: final results from long-term extension study and integrated database. Ann Rheum Dis. 2022 Mar;81(3):335-343. doi: 10.1136/annrheumdis-2021-221276. Epub 2021 Oct 27. PMID 34706874
- [Derived] Combe B, Balsa A, Sarzi-Puttini P, Tony HP, de la Torre I, Rogai V, Durand F, Witt S, Zhong J, Dougados M. Efficacy and safety data based on historical or pre-existing conditions at baseline for patients with active rheumatoid arthritis who were treated with baricitinib. Ann Rheum Dis. 2019 Aug;78(8):1135-1138. doi: 10.1136/annrheumdis-2018-214261. Epub 2019 Mar 6. No abstract available. PMID 30842122
- [Derived] Taylor PC, Kremer JM, Emery P, Zuckerman SH, Ruotolo G, Zhong J, Chen L, Witt S, Saifan C, Kurzawa M, Otvos JD, Connelly MA, Macias WL, Schlichting DE, Rooney TP, de Bono S, McInnes IB. Lipid profile and effect of statin treatment in pooled phase II and phase III baricitinib studies. Ann Rheum Dis. 2018 Jul;77(7):988-995. doi: 10.1136/annrheumdis-2017-212461. Epub 2018 Feb 20. PMID 29463520

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population included participants diagnosed with RA who had failed to respond adequately to any DMARD therapy, including biologics.
Pre-assignment Details: The study was divided into 3 distinct phases: Screening Phase (up to 28 days before randomization), Treatment Phase (12 weeks + 12-week extension period), and the Follow-up (4 ± 1 weeks following final dose of study medication).
Groups:
- Placebo: INCB028050 was administered once daily (QD), orally in matching placebo capsules. All participants were treated with only 1 capsule daily, without regard to meal time.
- Placebo Crossing Over to 7 mg INCB028050 QD: Participants that received placebo for the first 12 weeks were randomized to an active dosage of 7 mg INCB028050 QD.
- Placebo Crossing Over to 10 mg INCB028050 QD: Participants that received placebo for the first 12 weeks were randomized to an active dosage of 10 mg INCB028050 QD.
- INCB028050 4 mg QD: INCB028050 was administered qd, orally in 4 mg capsules. All participants were treated with only 1 capsule daily, without regard to meal time.
- INCB028050 7 mg QD: INCB028050 was administered qd, orally in 7 mg capsules. All participants were treated with only 1 capsule daily, without regard to meal time.
- INCB028050 10 mg QD: INCB028050 was administered qd, orally in 10 mg capsules. All participants were treated with only 1 capsule daily, without regard to meal time.
Period: Treatment Period (Weeks 0 Through 12)
Arm/Group | Placebo | Placebo Crossing Over to 7 mg INCB028050 QD | Placebo Crossing Over to 10 mg INCB028050 QD | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Started | 31 | 0 | 0 | 32 | 32 | 32
Safety Evaluable Participants | 31 | 0 | 0 | 31 | 32 | 31
Modified Intent-to-Treat Participants | 31 | 0 | 0 | 31 | 32 | 30
Completed (Participants completing Week 12) | 29 | 0 | 0 | 29 | 30 | 27
Not Completed | 2 | 0 | 0 | 3 | 2 | 5
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 1 | 2
Not completed — Consent Withdrawn | 1 | 0 | 0 | 0 | 0 | 2
Not completed — Protocol Deviation | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Not completed — corrected QT (QTc) exclusion criteria | 0 | 0 | 0 | 1 | 0 | 0
Period: Extension Period (Weeks 12 Through 24)
Arm/Group | Placebo | Placebo Crossing Over to 7 mg INCB028050 QD | Placebo Crossing Over to 10 mg INCB028050 QD | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Started | 0 | 14 | 15 | 29 | 30 | 27
Completed | 0 | 14 | 13 | 27 | 29 | 24
Not Completed | 0 | 0 | 2 | 2 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Consent Withdrawn | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Disease Progression | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0
Period: Follow-up (After Week 24)
Arm/Group | Placebo | Placebo Crossing Over to 7 mg INCB028050 QD | Placebo Crossing Over to 10 mg INCB028050 QD | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Started (Number of participants completed treatment) | 0 | 14 | 13 | 27 | 29 | 24
Safety Evaluable Participants (Population is inclusive of all safety participants continuing after Week 12.) | 0 | 14 | 15 | 29 | 30 | 27
Completed | 0 | 14 | 13 | 26 | 29 | 24
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: INCB028050 was administered qd, orally in matching placebo capsules. All participants were treated with only 1 capsule daily, without regard to meal time.
- Total: Total of all reporting groups
Arm/Group | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD | Placebo | Total
Number analyzed (Participants) | 32 | 32 | 32 | 31 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (12.28) | 53.7 (10.92) | 57.3 (10.38) | 55.2 (10.09) | 55.8 (10.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 25 | 22 | 102
  Male | 3 | 6 | 7 | 9 | 25

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Achieving American College of Rheumatology (ACR) 20 Improvement
Description: The ACR 20 is defined as ≥ 20% improvement in tender joint count plus ≥ 20% improvement in swollen joint count plus ≥ 20% improvement in 3 of the following 5 criteria: participants' assessment of pain, participants' global assessment of disease activity (PGA), Physician's global assessment of disease activity (PHGA), participants' self-assessed disability Health Assessment Questionnaire (HAQ), and Erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP), whichever shows the greatest change.
Time Frame: Week 12
Population: Modified Intent-to-Treat (mITT) population included all participants that enrolled, took at least 1 dose of study medication, and had both pre-dose and at least 1 post-baseline Rheumatoid arthritis (RA) assessment before Week 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 31 | 32 | 30
Participants | 10 | 16 | 19 | 16
Statistical Analysis 1: Comparison: Placebo vs INCB028050 4 mg QD vs INCB028050 7 mg QD vs INCB028050 10 mg QD; The prespecified primary analysis for ACR 20 was the Cochran-Armitage trend test looking for a dose-response relationship. The treatment effect was also assessed using a logistic regression model including background therapy (more than 8 weeks of biologics or not) and treatment; Test type: Superiority or Other; p = 0.0619, Cochran-Armitage trend test; Odds Ratio (OR) = 2.17, 95% CI 2-sided [0.77 to 6.15] — LOGISTIC regression model for odds ratio estimates : LOGIT(Response 0/1) = Treatment + Biologics
Statistical Analysis 2: Comparison: Placebo vs INCB028050 4 mg QD; Sensitivity analysis for pairwise comparisons of 4 mg QD versus placebo; Test type: Other; p = 0.1978, Fisher Exact
Statistical Analysis 3: Comparison: Placebo vs INCB028050 7 mg QD; Sensitivity analysis for pairwise comparisons of 7 mg QD versus placebo; Test type: Other; p = 0.0437, Fisher Exact
Statistical Analysis 4: Comparison: Placebo vs INCB028050 10 mg QD; Sensitivity analysis for pairwise comparisons of 10 mg QD versus placebo; Test type: Other; p = 0.1236, Fisher Exact

2. Primary Outcome: Participants With at Least 1 Adverse Event From Baseline Through Week 12
Time Frame: From Baseline through week 12
Population: Safety Evaluable Participants included all participants who were enrolled and took at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 31 | 32 | 31
Participants | 19 | 15 | 20 | 23

3. Secondary Outcome: Participants With at Least 1 Adverse Event From Week 12 to Week 24
Time Frame: Week 12 to Week 24
Population: Safety Evaluable Participants included all participants who were enrolled and took at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Crossing Over to 7 mg INCB028050 QD | Placebo Crossing Over to 10 mg INCB028050 QD | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 14 | 15 | 29 | 30 | 27
Participants | 6 | 5 | 12 | 16 | 16

4. Secondary Outcome: The Percentage of Participants Who Were Assigned to Active Treatment at Baseline Achieving ACR 20 Improvement at Week 24
Description: as for outcome 1
Time Frame: From Baseline to Week 24
Population: Modified Intent-to-Treat (mITT) population included all participants who were assigned to active treatment at baseline and had both pre-dose and at least 1 post-baseline Rheumatoid arthritis (RA) assessment before Week 12.
Measure: Count of Participants; unit: Participants
Arm/Group | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 27 | 30 | 25
Participants | 18 | 20 | 18

5. Secondary Outcome: The Percentage of Participants Achieving American College of Rheumatology (ACR) 50 Improvement at Week 12 and Week 24
Description: The ACR 50 is defined as ≥ 50% improvement in tender joint count plus ≥ 50% improvement in swollen joint count plus ≥50% improvement in 3 of the following 5 criteria: participants' assessment of pain, PGA, PHGA, participants' self-assessed disability HAQ, and ESR or CRP, whichever shows the greatest change.
Time Frame: Week 12 and Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 31 | 32 | 30
percentage of participants
  Week 12 | 13.0 | 35.0 | 31.0 | 30.0
  Week 24: number analyzed (Participants) | 31 | 27 | 30 | 25
  Week 24 | NA — Participants assigned to placebo either discontinued or crossed-over to active treatment at Week 12. | 33.0 | 37.0 | 44.0

6. Secondary Outcome: The Percentage of Participants Achieving American College of Rheumatology (ACR) 70 Improvement at Week 12 and Week 24
Description: The ACR 70 is defined as ≥ 70% improvement in tender joint count plus ≥ 70% improvement in swollen joint count plus ≥ 70% improvement in 3 of the following 5 criteria: participants' assessment of pain, PGA, PHGA, participants' self-assessed disability HAQ, and ESR or CRP, whichever shows the greatest change.
Time Frame: Week 12 and Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 31 | 32 | 30
percentage of participants
  Week 12 | 3.0 | 16.0 | 9.0 | 10.0
  Week 24: number analyzed (Participants) | 31 | 27 | 30 | 25
  Week 24 | NA — Participants assigned to placebo either discontinued or crossed-over to active treatment at Week 12. | 26.0 | 30.0 | 28.0

7. Secondary Outcome: The Percentage of Participants Achieving American College of Rheumatology (ACR) 90 Improvement at Week 12 and Week 24
Description: The ACR 90 is defined greater than or equal to (>=) 90 percent (%) improvement in painful and tender joint count; >= 90% improvement in swollen joint count; and >= 90% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP) at each visit.
Time Frame: Week 12 and Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 31 | 32 | 30
percentage of participants
  Week 12 | 0.0 | 3.0 | 0.0 | 3.0
  Week 24: number analyzed (Participants) | 31 | 27 | 30 | 25
  Week 24 | NA — Participants assigned to placebo either discontinued or crossed-over to active treatment at Week 12. | 11.0 | 10.0 | 12.0

8. Secondary Outcome: Change in Disease Activity Score 28 (DAS28) CRP Score From Baseline at Week 12 and Week 24
Description: Calculation of the disease activity score 28 (DAS 28) score was based on the tender joint count, plus swollen joint count, plus PGA, plus C-reactive protein (CRP). A higher score indicated more disease activity. The mean change from baseline (which represent decreases in the DAS 28 CRP scores) are shown as positive numbers in these analyses. The DAS28 provides a score on a scale from 0 to 10 indicating the current activity of the rheumatoid arthritis (>5.1=high disease activity; <3.2=low disease activity; <2.6=remission).
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 31 | 32 | 30
Units on a scale
  Baseline | 5.71 (0.875) | 5.64 (1.098) | 5.76 (0.925) | 5.64 (0.774)
  Change from baseline at Week 12 | -1.01 (1.245) | -1.87 (1.231) | -1.83 (1.534) | -1.84 (1.143)
  Change from baseline at Week 24: number analyzed (Participants) | 31 | 27 | 30 | 23
  Change from baseline at Week 24 | NA (NA) — Participants assigned to placebo either discontinued or crossed-over to active treatment at Week 12. | -2.13 (1.355) | -2.23 (1.548) | -2.75 (1.234)

9. Secondary Outcome: Change in Disease Activity Score 28 (DAS28) ESR Score From Baseline at Week 12 and Week 24
Description: Calculation of the disease activity score 28 (DAS 28) score was based on the tender joint count, plus swollen joint count, plus PGA, plus Erythrocyte sedimentation rate (ESR). The DAS28-ESR is expressed as units on a scale with the minimum score=0 (best) to maximum score=10 (worst). Remission was defined as DAS28-ESR <2.6. The mean change from baseline (which represent decreases in the DAS 28 ESR scores) are shown as positive numbers in these analyses.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 31 | 32 | 30
Units on a scale
  Baseline | 6.56 (0.840) | 6.41 (1.024) | 6.35 (0.968) | 6.37 (0.851)
  Change from baseline at Week 12 | -1.25 (1.489) | -1.87 (1.342) | -1.97 (1.613) | -1.90 (1.481)
  Change from baseline at Week 24: number analyzed (Participants) | 31 | 27 | 30 | 23
  Change from baseline at Week 24 | NA (NA) — Participants assigned to placebo either discontinued or crossed-over to active treatment at Week 12. | -2.17 (1.524) | -2.29 (1.455) | -2.79 (1.394)

10. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity by DAS28 (ESR)≤3.2
Description: Participants who achieved low disease activity based on the DAS 28 ESR (score ≤3.2). Participants who achieved low disease activity were classified as responders in this analysis.
Time Frame: Week 12 and Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 31 | 32 | 30
percentage of participants
  Week 12 | 19.0 | 23.0 | 31.0 | 13.0
  Week 24: number analyzed (Participants) | 31 | 27 | 30 | 23
  Week 24 | NA — Participants assigned to placebo either discontinued or crossed-over to active treatment at Week 12. | 48.0 | 53.0 | 65.0

11. Secondary Outcome: Percentage of Participants Achieving Remission by DAS28 (ESR) ≤2.6
Description: Participants who achieved inactive disease based on the DAS 28 ESR (score ≤2.6). Participants who achieved low disease activity were classified as responders in this analysis.
Time Frame: Week 12 and Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- Placebo to INCB028050 7 mg QD; Placebo to INCB028050 10 mg QD: Participants who were assigned to placebo group at baseline then crossed over to active treatment groups after week 12 were analyzed.
Arm/Group | Placebo to INCB028050 7 mg QD | Placebo to INCB028050 10 mg QD | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 15 | 16 | 31 | 32 | 30
percentage of participants
  Week 12 | 6.7 | 18.8 | 16.0 | 19.0 | 7.0
  Week 24: number analyzed (Participants) | 14 | 13 | 27 | 30 | 23
  Week 24 | 21.4 | 23.1 | 22.0 | 27.0 | 26.0

12. Secondary Outcome: Percentage of Participants Achieving Remission by DAS28 (CRP) ≤2.6
Description: Participants who achieved inactive disease based on DAS 28 CRP (score ≤2.6). Participants who achieved low disease activity were classified as responders in this analysis.
Time Frame: Week 12 and Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 32 | 30
percentage of participants
  Week 12 | 23.0 | 25.0 | 17.0
  Week 24: number analyzed (Participants) | 27 | 30 | 23
  Week 24 | 30.0 | 40.0 | 48.0

13. Secondary Outcome: Change in ACR Assessment Tender Joint Count (TJC) From Baseline to Week 12 and Week 24
Description: The 28 joints to be assessed for tenderness and swelling were shoulder, elbow, wrist, metacarpophalangeal (MCP) joints 1-5, proximal interphalangeal (PIP) joints 1-5, and knee on both sides of the body. The sum of tender joints ranged from 0 to 28 with 0 as best possible health status and 28 as worst health status.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Tender joints
Arm/Group | Placebo | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 31 | 32 | 30
Tender joints
  Baseline | 15.9 (6.67) | 14.4 (6.58) | 14.7 (6.70) | 15.9 (6.37)
  Change from baseline at Week 12 | -5.3 (6.40) | -7.4 (6.21) | -6.4 (7.98) | -8.8 (8.86)
  Change from baseline at Week 24: number analyzed (Participants) | 31 | 27 | 30 | 25
  Change from baseline at Week 24 | NA (NA) — Participants assigned to placebo either discontinued or crossed-over to active treatment at Week 12. | -8.3 (6.17) | -8.7 (7.42) | -12.0 (8.19)

14. Secondary Outcome: Change in ACR Assessment Swollen Joint Count (SJC) From Baseline to Week 12 and Week 24
Description: as for outcome 13
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Swollen joints
Arm/Group | Placebo | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 31 | 32 | 30
Swollen joints
  Baseline | 11.0 (5.28) | 12.0 (5.48) | 10.6 (4.57) | 12.9 (5.12)
  Change from baseline at Week 12 | -3.7 (4.02) | -6.1 (4.43) | -5.4 (5.85) | -7.2 (5.57)
  Change from baseline at Week 24: number analyzed (Participants) | 31 | 27 | 30 | 25
  Change from baseline at Week 24 | NA (NA) — Participants assigned to placebo either discontinued or crossed-over to active treatment at Week 12. | -7.3 (5.14) | -6.2 (5.04) | -9.1 (5.10)

15. Secondary Outcome: Change in Participants' Assessment of Pain From Baseline at Week 12 and Week 24
Description: Participants were to assess their current level of pain on a 100 mm horizontal Visual Analog Scale (VAS). The left-hand extreme of the line (0 mm) was described as "no pain" and the right-hand (100 mm) as "most imaginable pain".
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Placebo | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 31 | 32 | 30
millimeter (mm)
  Baseline | 62.37 (21.079) | 57.08 (24.716) | 63.25 (18.656) | 57.00 (22.995)
  Change from baseline at Week 12 | -6.24 (22.065) | -21.98 (26.275) | -22.19 (25.631) | -22.97 (37.691)
  Change from baseline at Week 24: number analyzed (Participants) | 31 | 27 | 30 | 25
  Change from baseline at Week 24 | NA (NA) — Participants assigned to placebo either discontinued or crossed-over to active treatment at Week 12. | -22.13 (27.294) | -27.62 (25.015) | -30.39 (30.847)

16. Secondary Outcome: Change in Participants' Global Assessment of Disease Activity From Baseline at Week 12 and Week 24
Description: Participants were to assess the disease (RA) activity on a 100 mm horizontal VAS. The left-hand extreme of the line (0 mm) was described as "no arthritis activity" (symptom-free and no arthritis symptoms) and the right hand extreme (100 mm) as "extremely active arthritis" (maximum arthritis disease activity). A decreasing mean score, therefore, indicates improvement.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Placebo | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 31 | 32 | 30
millimeter (mm)
  Baseline | 66.19 (20.522) | 59.02 (26.314) | 69.69 (18.893) | 62.25 (21.346)
  Change from baseline at Week 12 | -8.61 (22.569) | -22.06 (27.366) | -27.41 (21.990) | -25.48 (32.879)
  Change from baseline at Week 24: number analyzed (Participants) | 31 | 27 | 30 | 25
  Change from baseline at Week 24 | NA (NA) — Participants assigned to placebo either discontinued or crossed-over to active treatment at Week 12. | -24.02 (26.921) | -31.53 (23.891) | -34.08 (27.518)

17. Secondary Outcome: Change in Physician's Global Assessment of Disease Activity (PGA) From Baseline at Week 12 and Week 24
Description: Physicians were to assess the disease (RA) activity on a 100 mm horizontal VAS. The left-hand extreme of the line (0 mm) was described as "no arthritis activity" (symptom-free and no arthritis symptoms) and the right hand extreme (100 mm) as "extremely active arthritis" (maximum arthritis disease activity). A decreasing mean score, therefore, indicates improvement.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Placebo | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 31 | 32 | 30
millimeter (mm)
  Baseline | 63.45 (16.903) | 61.94 (19.162) | 59.80 (17.185) | 59.32 (16.890)
  Change from baseline at Week 12 | -20.23 (19.824) | -33.87 (24.283) | -29.95 (25.741) | -30.88 (19.334)
  Change from baseline at Week 24: number analyzed (Participants) | 31 | 27 | 30 | 25
  Change from baseline at Week 24 | NA (NA) — Participants assigned to placebo either discontinued or crossed-over to active treatment at Week 12. | -38.78 (22.527) | -36.94 (21.235) | -38.94 (21.776)

18. Secondary Outcome: Change in Health Assessment Questionnaire-Disability Index (HAQ-DI) From Baseline at Week 12 and Week 24
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 31 | 32 | 30
Score on a scale
  Baseline | 1.61 (0.494) | 1.50 (0.601) | 1.67 (0.474) | 1.50 (0.590)
  Change from baseline at Week 12 (n=31, 31, 30, 30) | -0.20 (0.367) | -0.38 (0.568) | -0.48 (0.613) | -0.33 (0.539)
  Change from baseline at Week 24: number analyzed (Participants) | 31 | 27 | 28 | 25
  Change from baseline at Week 24 | NA (NA) — Participants assigned to placebo either discontinued or crossed-over to active treatment at Week 12. | -0.56 (0.673) | -0.63 (0.563) | -0.39 (0.469)

19. Secondary Outcome: Change in Erythrocyte Sedimentation Rate (ESR) From Baseline at Week 12 and Week 24
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 millimeter/hour (mm/hr). A higher rate is consistent with inflammation.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Placebo | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 31 | 32 | 30
mm/hr
  Baseline | 40.8 (15.40) | 42.8 (17.62) | 37.3 (21.56) | 34.8 (29.05)
  Change from baseline at Week 12 | -6.1 (15.76) | -7.5 (23.17) | -10.7 (21.52) | -5.9 (32.35)
  Change from baseline at Week 24: number analyzed (Participants) | 31 | 27 | 30 | 23
  Change from baseline at Week 24 | NA (NA) — Participants assigned to placebo either discontinued or crossed-over to active treatment at Week 12. | -11.5 (21.96) | -12.8 (20.74) | -11.1 (26.00)

20. Secondary Outcome: Change in C-reactive Protein (CRP) From Baseline at Week 12 and Week 24
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 31 | 32 | 30
mg/L
  Baseline | 10.89 (11.556) | 15.63 (17.327) | 15.64 (16.113) | 7.52 (8.581)
  Change from baseline at Week 12 | 0.18 (10.063) | -9.76 (16.053) | -4.01 (26.799) | -0.73 (13.488)
  Change from baseline at Week 24: number analyzed (Participants) | 31 | 27 | 30 | 25
  Change from baseline at Week 24 | NA (NA) — Participants assigned to placebo either discontinued or crossed-over to active treatment at Week 12. | -6.74 (18.086) | -7.90 (16.713) | -5.52 (9.017)

21. Secondary Outcome: Change in Duration of Morning Stiffness From Baseline at Week 12 and Week 24
Description: Duration of morning stiffness was defined as the time elapsed when participant woke up in the morning and was able to resume normal activities without stiffness in minutes (If none was present = 0; If morning stiffness was continuing at the time of assessment or was unusual compared to the recent past, average of duration of stiffness over the past 3 days was reported; If stiffness persisted the entire day, 1440 minutes was recorded).
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 31 | 32 | 30
Minutes
  Baseline | 78.5 (61.36) | 179.8 (347.48) | 125.5 (246.75) | 79.2 (56.83)
  Change from baseline at Week 12 | 2.6 (69.23) | -51.1 (94.80) | -92.6 (250.51) | -42.2 (63.97)
  Change from baseline at Week 24: number analyzed (Participants) | 31 | 27 | 30 | 25
  Change from baseline at Week 24 | NA (NA) — Participants assigned to placebo either discontinued or crossed-over to active treatment at Week 12. | -120.6 (245.35) | -99.3 (254.05) | -51.5 (70.84)

22. Secondary Outcome: Percentage of Participants Achieving Good European League Against Rheumatism (EULAR) Response (DAS28 ESR) at Week 12
Description: EULAR response reflects an improvement in disease activity and an attainment of a lower degree of disease activity based on the DAS-28 score. A Good Response is defined as an improvement (decrease) in the DAS28 of more than 1.2 compared with Baseline and attainment of a DAS28 score less than or equal to 3.2.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 31 | 32 | 30
percentage of participants | 19.0 | 23.0 | 31.0 | 13.0

23. Secondary Outcome: Percentage of Participants Achieving Good EULAR Response (DAS28ESR) at Week 24
Description: as for outcome 22
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to INCB028050 7 mg QD | Placebo to INCB028050 10 mg QD | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 15 | 16 | 27 | 30 | 23
percentage of participants | 21.0 | 15.0 | 33.0 | 43.0 | 39.0

24. Secondary Outcome: Percentage of Participants Achieving Good EULAR Response (DAS28CRP) at Week 12
Description: EULAR response reflects an improvement in disease activity and an attainment of a lower degree of disease activity based on the DAS-28 score. A Good Response is defined as an improvement (decrease) in the DAS28 of more than 1.2 compared with Baseline and attainment of a DAS28 score less than or equal to 2.6.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 31 | 32 | 30
percentage of participants | 26.0 | 39.0 | 34.0 | 33.0

25. Secondary Outcome: Percentage of Participants Achieving Good EULAR Response (DAS28CRP) at Week 24
Description: as for outcome 24
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 27 | 30 | 23
percentage of participants | 48.0 | 53.0 | 65.0

26. Secondary Outcome: Change in SF-36 Mental Component Summary From Baseline at Week 12 and Week 24
Description: The Health Assessment Questionnaire Short Form 36 (SF-36) determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Scales 5-8 primarily contribute to the mental component summary score (PCS) of the SF-36. Scores on each scale are summed and averaged (range = 0 "worst"-100 "best").
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 31 | 32 | 30
scores on a scale
  Baseline | 71.08 (27.534) | 69.03 (28.181) | 78.41 (30.329) | 78.62 (24.160)
  Change from baseline at Week 12 | 2.92 (19.613) | 7.87 (19.547) | 2.21 (17.814) | 6.36 (25.203)
  Change from baseline at Week 24: number analyzed (Participants) | 31 | 27 | 30 | 25
  Change from baseline at Week 24 | NA (NA) — Participants assigned to placebo either discontinued or crossed-over to active treatment at Week 12. | 7.72 (17.543) | 4.60 (17.146) | 2.29 (28.869)

27. Secondary Outcome: Change in SF-36 Physical Component Summary From Baseline at Week 12 and Week 24
Description: The Health Assessment Questionnaire Short Form 36 (SF-36) determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Scales 1-4 primarily contribute to the physical component summary score (PCS) of the SF-36. Scores on each scale are summed and averaged (range = 0 "worst"-100 "best").
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 31 | 32 | 30
scores on a scale
  Baseline | 29.14 (14.330) | 34.67 (16.006) | 26.71 (14.642) | 28.82 (14.212)
  Change from baseline at Week 12 | 3.72 (11.027) | 9.57 (14.960) | 12.97 (17.932) | 8.35 (13.947)
  Change from baseline at Week 24: number analyzed (Participants) | 31 | 27 | 30 | 25
  Change from baseline at Week 24 | NA (NA) — Participants assigned to placebo either discontinued or crossed-over to active treatment at Week 12. | 11.60 (14.503) | 15.56 (16.144) | 11.77 (13.387)

28. Secondary Outcome: Percent of Participants Achieving a Minimum Clinically Important Difference (MCID) in the Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 12 and Week 24
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty. The MCID score for HAQ-DI is -0.22.
Time Frame: Week 12 and Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 31 | 32 | 30
percentage of participants
  Week 12 (n=31, 31, 30, 30) | 45.0 | 61.0 | 63.0 | 43.0
  Week 24: number analyzed (Participants) | 31 | 27 | 28 | 25
  Week 24 | NA — Participants assigned to placebo either discontinued or crossed-over to active treatment at Week 12. | 67.0 | 75.0 | 60.0

29. Secondary Outcome: Percent of Participants Achieving a MCID in the Pain Score (Participant's Assessment of Pain) at Week 12 and Week 24
Description: Participants were to assess their current level of pain on a 100 mm horizontal VAS. The left-hand extreme of the line (0 mm) was described as "no pain" and the right-hand (100 mm) as "most imaginable pain". MCID for the pain score is a decrease of at least 10 mm on a 100 mm scale.
Time Frame: Week 12 and Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 31 | 32 | 30
percentage of participants
  Week 12 | 35.0 | 58.0 | 69.0 | 67.0
  Week 24: number analyzed (Participants) | 31 | 27 | 30 | 25
  Week 24 | NA — Participants assigned to placebo either discontinued or crossed-over to active treatment at Week 12. | 59.0 | 70.0 | 72.0

30. Secondary Outcome: Percent of Participants Achieving a MCID in the SF-36 Physical Components and Mental Components at Week 12 and Week 24
Description: as for outcome 26
Time Frame: Week 12 and Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | INCB028050 4 mg QD | INCB028050 7 mg QD | INCB028050 10 mg QD
Number analyzed (Participants) | 31 | 31 | 32 | 30
percentage of participants
  Week 12 Physical Components | 52.0 | 68.0 | 69.0 | 57.0
  Week 24 Physical Components: number analyzed (Participants) | 31 | 27 | 30 | 25
  Week 24 Physical Components | NA — Participants assigned to placebo either discontinued or crossed-over to active treatment at Week 12. | 67.0 | 77.0 | 76.0
  Week 12 Mental Components | 52.0 | 58.0 | 41.0 | 50.0
  Week 24 Mental Components: number analyzed (Participants) | 31 | 27 | 30 | 25
  Week 24 Mental Components | NA — Participants assigned to placebo either discontinued or crossed-over to active treatment at Week 12. | 63.0 | 57.0 | 52.0

ADVERSE EVENTS:
Time Frame: Screening through follow-up visit up to approximately 8 months.
Description: Safety evaluable population included all randomized participants who received at least 1 dose of study drug. Those participants that continued after week 24 were safety subjects who continued after week 12.
  The data presented has been expanded to best represent the number at risk based on the dose and the period in which it was given to the participant.
Groups:
- Placebo (Weeks 0-12): INCB028050 was administered qd, orally in matching placebo capsules. All participants were treated with only 1 capsule daily, without regard to meal time.
- INCB028050 4 mg QD (Weeks 0-12): INCB028050 was administered qd, orally in 4 mg capsules. All participants were treated with only 1 capsule daily, without regard to meal time.
- INCB028050 7 mg QD (Weeks 0-12): INCB028050 was administered qd, orally in 7 mg capsules. All participants were treated with only 1 capsule daily, without regard to meal time.
- INCB028050 10 mg QD (Weeks 0-12): INCB028050 was administered qd, orally in 10 mg capsules. All participants were treated with only 1 capsule daily, without regard to meal time.
- Placebo to INCB028050 7 mg QD; Placebo to INCB028050 10 mg QD: 12-week extension period. Participants who were assigned to placebo group at baseline then crossed over to active treatment groups after week 12.
- INCB028050 4 mg QD (Weeks 12-24); INCB028050 7 mg QD (Weeks 12-24); INCB028050 10 mg QD (Weeks 12-24): 12-week extension period
- Placebo to INCB028050 7 mg QD (After Week 24 to Week 28); Placebo to INCB028050 10 mg QD (After Week 24 to Week 28): Follow-up Participants who were assigned to placebo group at baseline then crossed over to active treatment groups after week 12.
- INCB028050 4 mg QD (After Week 24 to Week 28); INCB028050 7 mg QD (After Week 24 to Week 28); INCB028050 10 mg QD (After Week 24 to Week 28): Follow-up
Arm/Group | Placebo (Weeks 0-12) | INCB028050 4 mg QD (Weeks 0-12) | INCB028050 7 mg QD (Weeks 0-12) | INCB028050 10 mg QD (Weeks 0-12) | Placebo to INCB028050 7 mg QD | Placebo to INCB028050 10 mg QD | INCB028050 4 mg QD (Weeks 12-24) | INCB028050 7 mg QD (Weeks 12-24) | INCB028050 10 mg QD (Weeks 12-24) | Placebo to INCB028050 7 mg QD (After Week 24 to Week 28) | Placebo to INCB028050 10 mg QD (After Week 24 to Week 28) | INCB028050 4 mg QD (After Week 24 to Week 28) | INCB028050 7 mg QD (After Week 24 to Week 28) | INCB028050 10 mg QD (After Week 24 to Week 28)
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 1/32 | 0/31 | 0/14 | 0/15 | 0/29 | 1/30 | 0/27 | 0/14 | 1/15 | 0/29 | 0/30 | 0/27
Other Adverse Events (participants affected / at risk) | 23/31 | 19/31 | 15/32 | 20/31 | 11/14 | 9/15 | 11/29 | 17/30 | 6/27 | 0/14 | 1/15 | 3/29 | 5/30 | 2/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Weeks 0-12) (N=31) | INCB028050 4 mg QD (Weeks 0-12) (N=31) | INCB028050 7 mg QD (Weeks 0-12) (N=32) | INCB028050 10 mg QD (Weeks 0-12) (N=31) | Placebo to INCB028050 7 mg QD (N=14) | Placebo to INCB028050 10 mg QD (N=15) | INCB028050 4 mg QD (Weeks 12-24) (N=29) | INCB028050 7 mg QD (Weeks 12-24) (N=30) | INCB028050 10 mg QD (Weeks 12-24) (N=27) | Placebo to INCB028050 7 mg QD (After Week 24 to Week 28) (N=14) | Placebo to INCB028050 10 mg QD (After Week 24 to Week 28) (N=15) | INCB028050 4 mg QD (After Week 24 to Week 28) (N=29) | INCB028050 7 mg QD (After Week 24 to Week 28) (N=30) | INCB028050 10 mg QD (After Week 24 to Week 28) (N=27)
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Weeks 0-12) (N=31) | INCB028050 4 mg QD (Weeks 0-12) (N=31) | INCB028050 7 mg QD (Weeks 0-12) (N=32) | INCB028050 10 mg QD (Weeks 0-12) (N=31) | Placebo to INCB028050 7 mg QD (N=14) | Placebo to INCB028050 10 mg QD (N=15) | INCB028050 4 mg QD (Weeks 12-24) (N=29) | INCB028050 7 mg QD (Weeks 12-24) (N=30) | INCB028050 10 mg QD (Weeks 12-24) (N=27) | Placebo to INCB028050 7 mg QD (After Week 24 to Week 28) (N=14) | Placebo to INCB028050 10 mg QD (After Week 24 to Week 28) (N=15) | INCB028050 4 mg QD (After Week 24 to Week 28) (N=29) | INCB028050 7 mg QD (After Week 24 to Week 28) (N=30) | INCB028050 10 mg QD (After Week 24 to Week 28) (N=27)
Headache (Nervous system disorders) | 2 | 4 | 3 | 3 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 1 | 3 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 2 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study; provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.